CLINICAL TRIAL: NCT05270395
Title: Piloting 'mPal,' a Multilevel Implementation Strategy to Integrate Non-hospice Palliative Care Into Advanced Stage Lung Cancer Treatment
Brief Title: Piloting 'mPal,' a Multilevel Strategy for Palliative Care Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laurie McLouth (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Laurie McLouth, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 74152; 2KL2TR001996-05A1 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-03-08 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Palliative care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mPal intervention (Experimental): Participants in this group will receive the mPal intervention. mPal's patient content includes a multi-component web-based tool with the following: (1) a brief educational video that seeks to educate patients about palliative care; (2) and assessment of palliative care knowledge; (3) assessment of palliative care needs; and (4) an assessment of whether patients would like to meet with palliative care or discuss palliative care and their palliative care needs with their oncology provider. mPal's provider content (not randomized) will include education. System-level modifications will also be made to the electronic health record to facilitate palliative care discussions and referrals.
  Interventions: Behavioral: mPal
- Standard of care (No Intervention): Participants in this group will receive standard of care (applies to patients only).

INTERVENTIONS:
Behavioral: mPal — mPal's patient content includes a multi-component web-based tool with the following: (1) a brief educational video that seeks to educate patients about palliative care; (2) and assessment of palliative care knowledge; (3) assessment of palliative care needs; and (4) an assessment of whether patients would like to meet with palliative care or discuss palliative care and their palliative care needs with their oncology provider.
  The provider-level component includes provider education on palliative care. The system-level component includes electronic health record modifications to facilitate palliative care discussions and referrals.
  Arms: mPal intervention

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of mPal, a multilevel implementation strategy to improve palliative care use among advanced stage lung cancer patients receiving cancer treatment.

DETAILED DESCRIPTION:
In this study, 60 advanced stage lung cancer patients will be randomized to mPal's patient-level component or usual care. Oncology providers will receive the mPal intervention. mPal is designed to help oncology providers integrate outpatient palliative care (non-hospice palliative care; NHPC) into routine clinical practice through: 1) electronic health record enhancements; 2) patient education and preparation for NHPC discussions when patients are in clinic to see their oncology providers; and 3) provider education about NHPC.

This study will examine the feasibility and acceptability of mPal and gather preliminary data on potential outcomes for a future effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* new or recurrent AJCC stage IIIb-IV non-small cell lung cancer or extensive stage small cell lung cancer
* ECOG performance status 0-3/Karnofsky 40-100
* at least three weeks into active oncologic treatment (chemotherapy, immunotherapy, chemo-immunotherapy)

Exclusion Criteria:

* unstable brain metastases
* Cognitive (i.e., dementia) or psychiatric condition (e.g., psychotic disorder) for which participating would be inappropriate
* Receiving palliative care
* Unable to speak and read English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie McLouth, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, individuals were not randomized until they completed the baseline assessment. Although 75 participants were consented, only 68 completed baseline assessments and were randomized.
Groups:
- mPal Intervention: Participants in this group will receive the mPal intervention. mPal's patient content includes a multi-component web-based tool with the following: (1) a brief educational video that seeks to educate patients about palliative care; (2) and assessment of palliative care knowledge; (3) assessment of palliative care needs; and (4) an assessment of whether patients would like to meet with palliative care or discuss palliative care and their palliative care needs with their oncology provider. mPal's provider content (not randomized) will include education. System-level modifications will also be made to the electronic health record to facilitate palliative care discussions and referrals.
  mPal: mPal's patient content includes a multi-component web-based tool with the following: (1) a brief educational video that seeks to educate patients about palliative care; (2) and assessment of palliative care knowledge; (3) assessment of palliative care needs; and (4) an assessment of whether patients would like to meet with palliative care or discuss palliative care and their palliative care needs with their oncology provider.
  The provider-level component includes provider education on palliative care. The system-level component includes electronic health record modifications to facilitate palliative care discussions and referrals.
Period: Overall Study
Arm/Group | mPal Intervention | Standard of Care
Started | 34 | 34
Completed | 30 | 30
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 1 | 2
Not completed — Study Team Withdrew | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mPal Intervention | Standard of Care | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.3) | 61.0 (11.5) | 62.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 31 | 64
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 29 | 28 | 57
  More than one race | 1 | 0 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment
Description: Enrollment feasibility is defined as the number of eligible and approached patients who agree to participate
Time Frame: up to 6 months
Population: Participants were not randomized until they completed baseline assessment, thus, this number is the total individuals eligible.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Participants eligible for study and approached to join study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 118
Participants | 75

2. Secondary Outcome: Patient Palliative Care Referrals
Description: Number of patients in each arm who receive a referral to palliative care within 1-month and 3-months post-intervention
Time Frame: up to 3-months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 34 | 34
Participants | 2 | 2

3. Secondary Outcome: Acceptability of Intervention
Description: 4-item acceptability of intervention measure (AIM); items responded to on a 5-point Likert-type scale (1 - 5) with higher scores indicating greater acceptability.
Time Frame: up to 2 weeks post-intervention viewing
Population: The intervention was only administered to the mPal arm. Participants that completed enough items to calculate a score were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 31 | 0
score on a scale | 3.95 (0.64) |

4. Secondary Outcome: Change in Palliative Care Attitudes
Description: Palliative Care Attitudes Scale; 9-items responded to on a Likert-type scale (range 9 - 60) with higher scores indicating more favorable attitudes and motivation towards palliative care. Mean change in total score at Time 2 is presented, adjusted for the baseline value of PCAS Total Score at baseline, age, and sex.
Time Frame: Baseline, up to 2-months post intervention
Population: Participants that completed enough items at the Time 2 assessment were included in the analysis
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 28
score on a scale | 1.12 (1.33) | -0.07 (1.37)

5. Secondary Outcome: Feasibility of Intervention
Description: 4-item feasibility of intervention measure (FIM); items responded to on a 5-point Likert-type scale (1 - 5) with higher scores indicating higher feasibility.
Time Frame: up to 2 weeks post-intervention viewing
Population: Administered only to intervention participants; Participants that completed enough items at the Time 2 assessment were included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 31 | 0
score on a scale | 4.03 (0.56) |

6. Secondary Outcome: Feasibility of Retention
Description: Feasibility of retention is defined as the number of patients who complete baseline and follow-up questionnaire
Time Frame: up to 2-months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 34 | 34
Participants | 30 | 30

7. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 1: How Would You Describe Your Level of Knowledge About Palliative Care?
Description: The percentage of participants responding, "know what palliative care is and could explain it to someone else" reported. Odds ratio was calculated using logistic regression.
  Item 1 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to respond to this question: "How would you describe your level of knowledge about palliative care?" Participants can respond, "I've never heard of it," "I know a little bit about palliative care," or "I know what palliative care is and could explain it to someone else."
  For the analysis, the first two responses were collapsed to create a dichotomous variable ("have no or little knowledge of palliative care" versus "know what palliative care is and could explain it to someone else").
Time Frame: Baseline and at 1-month follow-up
Population: We analyzed all available cases at Time 2 assessment, which included participants that completed enough items to be included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 28 | 28
Percentage of participants | 35.71 | 14.29
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; We conducted logistic regression to predict knowledge of palliative care (as measured by ten items in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire) in the mPal intervention arm and in the standard of care arm at 1-month post-intervention, adjusting for baseline value of each item, age, and sex; Test type: Superiority; p = 0.02, Regression, Logistic; Odds Ratio (OR) = 8.02, 95% CI 2-sided [1.38 to 46.69]

8. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 2: Help Friends and Family to Cope With a Patient's Illness
Description: The percentage of participants responding, "Agree" reported. Odds ratio was calculated using logistic regression.
  Item 2 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement regarding the goal of palliative care: "Help friends and family to cope with a patient's illness." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree" ("Strongly agree" or "Somewhat agree") versus "Disagree/Don't know" ("Somewhat disagree," "Strongly disagree," or "Don't know"). For this item, "Agree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 27
Percentage of participants | 76.67 | 70.37
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.63, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.40 to 4.56]

9. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 3: Offer Social and Emotional Support
Description: The percentage of participants responding, "Agree" reported. Odds ratio was calculated using logistic regression.
  Item 3 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement regarding the goal of palliative care: "Offer social and emotional support." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree" ("Strongly agree" or "Somewhat agree") versus "Disagree/Don't know" ("Somewhat disagree," "Strongly disagree," or "Don't know"). For this item, "Agree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 26
Percentage of participants | 73.33 | 88.46
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.13, Regression, Logistic; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.06 to 1.46]

10. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 4: Manage Pain and Other Physical Symptoms
Description: The percentage of participants responding, "Agree" reported. Odds ratio was calculated using logistic regression.
  Item 4 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement regarding the goal of palliative care: "Manage pain and other physical symptoms." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree" ("Strongly agree" or "Somewhat agree") versus "Disagree/Don't know" ("Somewhat disagree," "Strongly disagree," or "Don't know"). For this item, "Agree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 26
Percentage of participants | 76.67 | 84.62
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.40, Regression, Logistic; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.13 to 2.24]

11. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 5: Give Patients More Time at the End of Life
Description: The percentage of participants responding, "Disagree" reported. Odds ratio was calculated using logistic regression.
  Item 5 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement regarding the goal of palliative care: "Give patients more time at the end of life." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree/Don't know" ("Strongly agree," "Somewhat agree," or "Don't know") versus "Disagree" ("Somewhat disagree" or "Strongly disagree"). For this item, "Disagree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 26
Percentage of participants | 26.67 | 15.38
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.51 to 9.62]

12. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 6: Accepting Palliative Care Means Giving up
Description: The percentage of participants responding, "Disagree" reported. Odds ratio was calculated using logistic regression.
  Item 6 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement about palliative care: "Accepting palliative care means giving up." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree/Don't know" ("Strongly agree," "Somewhat agree," or "Don't know") versus "Disagree" ("Somewhat disagree" or "Strongly disagree"). For this item, "Disagree" signified positive belief about palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 27
Percentage of participants | 80.00 | 62.96
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 3.55, 95% CI 2-sided [0.88 to 14.32]

13. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 7: It is a Doctor's Obligation to Inform All Patients With Cancer About the Option of Palliative Care
Description: The percentage of participants responding, "Agree" reported. Odds ratio was calculated using logistic regression.
  Item 7 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement about palliative care: "It is a doctor's obligation to inform all patients with cancer about the option of palliative care." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree" ("Strongly agree" or "Somewhat agree") versus "Disagree/Don't know" ("Somewhat disagree," "Strongly disagree," or "Don't know"). For this item, "Agree" signified positive belief about palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 29 | 28
Percentage of participants | 72.41 | 67.86
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.09, Regression, Logistic; Odds Ratio (OR) = 3.93, 95% CI 2-sided [0.82 to 18.89]

14. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 8: If You Accept Palliative Care, You Must Stop Other Treatments
Description: The percentage of participants responding, "Disagree" reported. Odds ratio was calculated using logistic regression.
  Item 8 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement about palliative care: "If you accept palliative care, you must stop other treatments." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree/Don't know" ("Strongly agree," "Somewhat agree," or "Don't know") versus "Disagree" ("Somewhat disagree" or "Strongly disagree"). For this item, "Disagree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 27
Percentage of participants | 73.33 | 62.96
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.42, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.46 to 6.43]

15. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 9: Palliative Care is the Same as Hospice Care
Description: The percentage of participants responding, "Disagree" reported. Odds ratio was calculated using logistic regression.
  Item 9 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement about palliative care: "Palliative care is the same as hospice care." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree/Don't know" ("Strongly agree," "Somewhat agree," or "Don't know") versus "Disagree" ("Somewhat disagree" or "Strongly disagree"). For this item, "Disagree" signified correct knowledge of palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 27
Percentage of participants | 66.67 | 48.15
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 2.86, 95% CI 2-sided [0.87 to 9.42]

16. Secondary Outcome: Change in Palliative Care Knowledge - Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS), Item 10: When I Think of "Palliative Care," I Automatically Think of Death
Description: The percentage of participants responding, "Disagree" reported. Odds ratio was calculated using logistic regression.
  Item 10 in the Health Information National Trends Survey Palliative Care Knowledge and Perceptions Questionnaire (HINTS) asks participants to state the degree to which they agree or disagree with this statement about palliative care: "When I think of "palliative care," I automatically think of death." Participants can respond, "Strongly agree," "Somewhat agree," "Somewhat disagree," "Strongly disagree," or "Don't know."
  For the analysis, we dichotomized the responses into "Agree/Don't know" ("Strongly agree," "Somewhat agree," or "Don't know") versus "Disagree" ("Somewhat disagree" or "Strongly disagree"). For this item, "Disagree" signified positive belief about palliative care.
Time Frame: Baseline and at 1-month follow-up
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | mPal Intervention | Standard of Care
Number analyzed (Participants) | 30 | 26
Percentage of participants | 70.00 | 34.62
Statistical Analysis 1: Comparison: mPal Intervention vs Standard of Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 8.29, 95% CI 2-sided [1.99 to 34.49]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | mPal Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/34 | 2/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05270395/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT05270395/ICF_000.pdf